CLINICAL TRIAL: NCT05930574
Title: Demographic and Clinical Characterization of Patients Operated by the General Surgery Service Who Were Admitted by the Emergency Service of the Dr. Rafael Ángel Calderón Guardia Hospital, 2021-2022.
Brief Title: Implementation of an Epidemiological and Clinical Registry of Emergency Surgery Patients in a Costa Rican Hospital
Status: Completed | Type: Observational
Sponsor: Caja Costarricense de Seguro Social (Other Government)
Responsible Party: Principal Investigator, María Rosario Espinoza Mora, Head of the Health Investigation Department, Hospital Dr. Rafael Angel Calderón Guardia, Caja Costarricense de Seguro Social
Other Study IDs: 01-UIS-HCG-2023
Record Dates: First submitted 2023-06-24; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Surgical Complication; Emergencies
Keywords: Registry; Trauma; General surgery; Emergency
MeSH Terms: conditions — Emergencies; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Abdominal surgery — surgical interventions by gastrointestinal emergencies, hepatobiliary emergencies and trauma

SUMMARY:
A retrospective cross-sectional study was conducted in a quaternary level university hospital of the Costa Rican public health system. The study included all patients aged 12 years and older who required emergency surgery by the hospital's emergency surgery and trauma service, admitted through the hospital's emergency service.

DETAILED DESCRIPTION:
This research consists in a retrospective cross-sectional study carried out in a quarterly level university hospital of care of the Costa Rican public health system (high complexity). The study included all patients aged 12 years or older who required emergency surgery for the hospital's emergency surgery and trauma service, admitted to this center between 2020 and 2022. Only those patients who required emergency surgery by another surgical specialty during this period were excluded from the register. A non-probabilistic convenience sampling was performed, based on the pre-established selection criteria and determined by the number of patients treated in the shock room of the hospital, that subsequently received general emergency or trauma surgery in the period under study. Sociodemographic variables, hemodynamic status, period of hospitalization, related to the procedure performed and the underlying comorbidities, as well as the clinical outcome, were included in the study database.

ELIGIBILITY:
Inclusion Criteria:

* The study included all patients aged 12 years and older who required emergency surgery by the hospital's emergency surgery and trauma service, admitted through the hospital's emergency service.

Exclusion Criteria:

* . Only those patients who required emergency surgery by another surgical specialty during this period were excluded from the register.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring emergency surgery by the hospital's emergency surgery and trauma service, admitted through the hospital's emergency service.
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | retrospective study (2020-2022)
  Mortality rate after the surgical procedure during hospitalization
Mechanical ventilation | retrospective study (2020-2022)
  Days of mechanical ventilation needed
Requirement of Intensive Care Unit | retrospective study (2020-2022)
  Days of permanence in Intensive Care Unit
Infections | retrospective study (2020-2022)
  Infection rate after the surgical procedure during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investigación en Salud, Hospital Dr. Rafael Angel Calderón Guardia, San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No
The public health system of Costa Rica avoid sharing clinical data with external centers.